CLINICAL TRIAL: NCT06491264
Title: Concurrent Multiparameter Optimized Noninvasive Brain Stimulation for Working Memory in Aging
Brief Title: Multiparameter Optimized tES for Memory in Aging
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Kevin Caulfield, Assistant Professor, Medical University of South Carolina
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00133951
Record Dates: First submitted 2024-04-17; First posted 2024-07-09 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-01

CONDITIONS: Healthy Aging
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: In this within-subjects design, participants will each receive 5 sessions of tES in a counterbalanced order. tES will be applied using different stimulation intensities that are personalized to each person using MRI scans. tES will also have different 4 different waveforms (theta, gamma, theta-gamma ranges or none).
Who Masked: Participant, Investigator
Masking Description: Double-blind, sham-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- Personalized tES stimulation #1 (Experimental): tES will be applied with personalized parameters in condition #1 for approximately 20 minutes.
  Interventions: Device: Transcranial electrical stimulation
- Personalized tES stimulation #2 (Experimental): tES will be applied with personalized parameters in condition #2 for approximately 20 minutes.
  Interventions: Device: Transcranial electrical stimulation
- Personalized tES stimulation #3 (Experimental): tES will be applied with personalized parameters in condition #3 for approximately 20 minutes.
  Interventions: Device: Transcranial electrical stimulation
- Standard tES (Experimental): Standard tES will be applied in condition #4 for approximately 20 minutes.
  Interventions: Device: Transcranial electrical stimulation
- Sham tES stimulation (Sham Comparator): A sham (placebo) comparison condition will be applied in condition #5 for approximately 20 minutes.
  Interventions: Device: Transcranial electrical stimulation

INTERVENTIONS:
Device: Transcranial electrical stimulation — We will administer active transcranial electrical stimulation in one of the 4 active stimulation conditions and 1 sham stimulation condition.

SUMMARY:
With an aging population worldwide, it is critical to develop effective interventions promoting healthy cognitive aging. Transcranial electrical stimulation (tES) is a promising but not fully realized noninvasive brain stimulation approach that could improve memory. This study investigates the behavioral and electrocortical effects of personalized tES in aging to determine whether whether optimal dosing, electrode placements, and waveforms elicit stronger responses.

DETAILED DESCRIPTION:
With an aging population worldwide, it is critical to develop effective interventions promoting healthy cognitive aging. A key component of healthy cognition is intact working memory, an executive neural process holding information temporarily. With increasing age, working memory capacity decreases and is associated with a loss of independence, thus incentivizing the need to retain a healthy working memory capacity. In addition to facilitating healthy aging, developing a method that improves working memory could help those diagnosed with mild cognitive impairment (MCI) and Alzheimer's Disease (AD), which is currently is the 6th leading cause of death in the US and has an annual economic burden of $305 billion.

A potential approach to improve working memory is transcranial electrical stimulation (tES), a noninvasive brain stimulation method using scalp electrodes to deliver low electrical currents of 2 milliamps (mA) over the cortical target. While some prior studies have shown that prefrontal tES can improve working memory in older adults, there are small meta-analytic effect sizes and no FDA-approved indications to date. These mixed results could be due to applying one-size-fits-all and suboptimal tES parameters. In this study, the investigators will test the effects of personalized parameters, including dosing, electrode positioning, and waveforms compared to standard tES and placebo.

ELIGIBILITY:
Inclusion Criteria:

* 50 - 85 y.o.
* Endorse good health with no history of mental or physical illness
* Willingness to adhere to the study schedule and assessments
* Able to read consent document and provide informed consent.
* English is a first or primary fluent language.

Exclusion Criteria:

* Any current psychiatric diagnosis or current Clinical Global Impression ratings of psychiatric illness > 1
* Neurodevelopmental disorders, history of Central Nervous System (CNS) disease, concussion, overnight hospitalization, or other neurologic sequela, tumors, seizures, meningitis, encephalitis, or abnormal CT or MRI of the brain
* Any psychotropic medication is taken within 5 half-lives of procedure time
* Any head trauma resulting in loss of consciousness
* Visual impairment (except the use of glasses)
* Inability to complete cognitive testing
* Active participation or plan for enrollment in another evidence-based clinical trial affecting the psychosocial function
* Repeated abuse or dependence upon drugs (excluding nicotine and caffeine) or taking medications including stimulants, modafinil, thyroid medication, or steroids
* Implanted devices/ferrous metal of any kind
* History of seizure or epilepsy, currently taking medications that lower seizure thresholds
* Claustrophobia or other conditions that would prevent the MRI assessment.
* Pregnancy (or suspected/possible pregnancy or plan to become pregnant in the short term).
* Urine Pregnancy Test: If the subject is a woman of childbearing potential and /or a man capable of fathering a child before, during, and/or after participation precautions should be taken. Examples of acceptable methods of birth control for participants involved in the study include birth control pills, patches, Intrauterine Devices (IUD), condoms, sponges, diaphragm with spermicide, or avoiding sexual activity that could cause the subject to become pregnant.
* Inability to adhere to the treatment schedule.
* Inability to fit the wearable device to the user's head.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Electrocortical EEG changes pre- to post-tES | 1 year
  Observe effects of each tES condition within each of the 5 sessions, as measured by TMS-EEG
N-back working memory changes pre- to post-tES | 1 year
  Observe effects of each tES condition within each of the 5 sessions on the N-back memory task

SECONDARY OUTCOMES:
Rate of side effects from tES | 1 year
  Questionnaire regarding headache, scalp sensation, and other common side effects of tES on a scale of 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Caulfield, PhD, Principal Investigator — Medical University of South Carolina

IPD SHARING:
Plan to Share IPD: No